CLINICAL TRIAL: NCT03095976
Title: Amnion-Chorion Allograft Barrier Used for Root Surface and Guided Tissue Regeneration for Periodontal Intrabony Defects and Grade II Furcation Defects.
Brief Title: Amnion-Chorion Allograft Barrier Used for Root Surface and Guided Tissue Regeneration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Yusuke Hamada, Clinical Assistant Professor, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1608175133
Record Dates: First submitted 2017-03-24; First posted 2017-03-30 (Actual); Results first posted 2021-04-14 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-03

CONDITIONS: Periodontal Diseases
Keywords: Guided Tissue Regeneration,; Amnion-Chorion,; Intrabony defects,; furcation
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Intervention Model Description: Prospective Case Series
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Test group (Experimental): Application of Amnion-Chorion allograft membrane (ACM) on the root surface of periodontally diseased teeth in conjunction with corticocancellous allograft bone substitute covered by ACM in a combination GTR treatment of periodontal intrabony and furcation defects.
  Interventions: Procedure: Amnion-Chorion allograft membrane on the root surface of periodontally diseased site.

INTERVENTIONS:
Procedure: Amnion-Chorion allograft membrane on the root surface of periodontally diseased site. — Application of Amnion-Chorion allograft membrane (ACM) on the root surface of periodontally diseased teeth in conjunction with corticocancellous allograft bone substitute covered by ACM in a combination GTR treatment of periodontal intrabony and furcation defects

SUMMARY:
The purpose of this pilot project is to evaluate the efficacy of application of Amnion-Chorion allograft membrane on the root surface of periodontally diseased teeth in conjunction with bone substitute covered by Amnion-Chorion allograft in a combination Guided Tissue Regeneration (GTR) treatment of periodontal intrabony and furcation defects.

DETAILED DESCRIPTION:
Patients who are referred to the Graduate Periodontics Clinic at Indiana University School of Dentistry for the treatment of severe chronic/aggressive periodontitis will be screened for possible participation in this study. Up to 20 subjects will be accepted into this study.

Written informed consent and authorization will be obtained from all participants and they will be given a copy of the signed informed consent documents.

The procedures listed below are all within standard care for a regenerative therapy around the teeth except the application of the membrane on the root surface prior to the bone grafting. No data collected for this study will be taken from sources outside of that already recorded for standard of care procedures.

Clinical Measurements A single calibrated examiner will perform clinical baseline and 6-month follow up measurements. O'Leary plaque score will be assessed. Six sites of each tooth of probing depth (PD), recession (REC) and clinical attachment level (CAL) will be recorded to the nearest millimeter with a University of North Carolina Probe (UNC Probe). For Glickman grade II furcation defects, in addition to the previous measurements, vertical probing pocket depth (VPD) and horizontal probing depth (HPD) will be measured.

Radiographic assessment will be performed with vertical bite-wing radiographs at baseline and 6-month post-surgical treatment. In order to maximize the standardization of the angulation of radiographs, bite registration will be taken prior to the first radiograph and utilized with beam-guiding device. It will be stored to be used post operatively. Sirona Dental Systems© with 7mA 60kV with 0.16s exposure time will be utilized for all radiographs. Digital #2 films manufactured by Air Techniques Inc. will be used for radiographic assessment. Bony defect (BD) will be defined as the most coronal point where the periodontal ligament space showed a continuous width. If several bony contours could be identified, the most apical one that crossed the root will be defined as the boney defect and the most coronal one as alveolar crest. If the cemento-enamel junction (CEJ) was destroyed by the restorative treatment, the margin of the restoration will be taken as a landmark. Beam guided device will be used as a calibration of measurements. The change of bone fill and angulation will be recorded.

All surgery will be rendered at the Graduate Periodontics Clinic at Indiana University School of Dentistry. All the patients will be treated under local anesthesia (2% lidocaine with 1/100,000epi or 4% articaine with 1/100,000epi). If the patient is willing to receive the surgery under intravenous or oral sedation, those services will be provided based on the necessity. After local anesthesia, intracrevicular incisions will be made and full-thickness mucoperiosteal flaps will be raised both buccally and lingually; the surgeon will try to preserve the maximum extent of the marginal and interdental gingival tissue to obtain primary closure and membrane coverage. Vertical releasing incisions will only be used if necessary to gain access for defect debridement. The alveolar bone will be exposed at least 3 mm beyond the edges of the defect, and periosteal releasing incisions will be made to ensure complete membrane coverage at the time of suturing if necessary. All granulation tissue will be removed, the defects will be debrided, and the roots will be thoroughly scaled and root planed by hand instruments and ultrasonic devices. Following debridement, 17% Ethylenediaminetetraacetic acid (EDTA) solution with cotton pellet will be applied on the root surface for 2 minutes. After thorough irrigation with saline, BioXclude® (Amnion-Chorion Membrane: Food and Drug Administration (FDA) Approved materials for intrabony defects) will be cut into two pieces. The amnion-chorion BioXclude membrane is regulated by the FDA under section 361 of the Public Health Service Act as a "Human cells, tissues, and cellular or tissue-based product" (HCT/P). The FDA does not require pre-market approval for these products like it would with drugs, biologics or devices. Therefore, this product will have no associated "investigational device exemption" (IDE) number. The FDA views using amnion chorion as a wound covering to aid in the healing of tissues throughout the body to be a "homologous use". One goes to the root surface, and coronal portion of the membrane has to be >3mm coronal of CEJ. Once applied the membrane, one drop of saline will be applied to obtain better adaptation of membrane on the root surface. Bone substitutes 0.5cc (Particle size of 0.25-0.5mm of Corticocancellous, Maxxeus®) will be hydrated for at least 10min prior to application, and applied into the defects. The bone particles will not exceed the edge of defects in order to avoid over fill. Following the bone graft will be delivered to the defect. The coronal portion of excessive membrane will be just folded over the graft materials. The other BioXclude membrane will be utilized over the grafts, and will always be placed coronal to the interproximal bone crest so that it completely covers the defect and extends 2 to 3 mm beyond the residual bone. No sutures, pins, or tacks will be used for membrane fixation or stabilization. The orientation of the membrane will not matter. Vertical or horizontal mattress sutures with 5-0 Proline (Monofilament/Nylon) will be placed in the interproximal tissues to obtain primary closure as much as possible.

Intra-surgical Clinical Measurements. Intrabony defects: defect morphology will be measured (1 wall, 2 walls and/or those combinations) from the deepest aspect of the defect from the most coronal side of edge of the defects.

Furcation defects: 1) Cementoenamel junction to roof of furcation (CEJ-ROF); 2) roof of furcation to base of defect (ROF-BOD); 3) roof of furcation to crest of bone at furcation entrance (ROF-COB); 4) crest of bone to base of defect (COB-BOD); 5) root divergence at crest of bone (RDCB); 6) horizontal extent (base) of defect at level of furcation entrance (HBODF); 7) horizontal extent (base) of defect at level of crest of bone (HBOD-C); and 8) cemento-enamel junction to interproximal crest of bone (CEJ-INTPRX)

All patients will receive antibiotics (875mg amoxicillin twice /day) for one week. If participants are allergic to amoxicillin, clindamycin (150mg twice/day) for one week will be prescribed. Analgesics (600mg ibuprofen three times/day) will be prescribed as needed for discomfort. Pt will be seen one, two and four weeks as a post-operative follow up. Patients will be advised to rinse twice daily with 0.12% chlorhexidine for 2 weeks after surgery. Patients will be instructed to refrain from brushing the teeth in the surgical area for 2 weeks. After that, they will be instructed to initiate brushing with an extra-soft toothbrush. Subjects will be recalled at 4-week intervals after 4weeks from surgical procedure for a period of 6 months for plaque scoring, oral hygiene instruction, and professional prophylaxis as needed. No subgingival probing or instrumentation will be performed at the experimental sites until the 6-month follow-up appointment.

ELIGIBILITY:
Inclusion Criteria:

1. ASA class I or II;
2. age >18 years old;
3. Non-smoker;
4. diagnosis of chronic or aggressive periodontitis previously treated with nonsurgical mechanical debridement; 5) patients have at least one two-wall intrabony defect in interproximal areas with radiographic evidence of an intrabony component of ≥ 4 mm, PPD ≥ 6 mm with 1-wall or 2-wall or combination of those defects;

6) Glickman Grade II furcation involvement on buccal of mandibular or maxillary first or second molars without soft tissue exposure of furcation entrance; 7) tooth mobility Miller Grade <1; 8) more than 2mm of keratinized tissue with those selected teeth.

Exclusion Criteria:

1. did not meet all inclusion criteria;
2. pregnancy or nursing woman;
3. subjects with active systemic or localized infection (exclude chronic periodontitis);
4. poor compliance or failure to maintain good oral hygiene as ascertained by the presence of full-mouth plaque score ≥ 20%;
5. restorations or caries on root surfaces or untreated endodontic infections;
6. participants received periodontal surgical treatment on the same site of this study within 2 years;
7. use of systemic or local antibiotics on the anticipated surgical sites during the past 3 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2017-06-14 (Actual); Primary Completion 2019-09-10 (Actual); Study Completion 2019-09-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University School of Dentistry, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Eke PI, Dye BA, Wei L, Thornton-Evans GO, Genco RJ; CDC Periodontal Disease Surveillance workgroup: James Beck (University of North Carolina, Chapel Hill, USA), Gordon Douglass (Past President, American Academy of Periodontology), Roy Page (University of Washin. Prevalence of periodontitis in adults in the United States: 2009 and 2010. J Dent Res. 2012 Oct;91(10):914-20. doi: 10.1177/0022034512457373. Epub 2012 Aug 30. PMID 22935673
- [Background] Bowers GM, Schallhorn RG, McClain PK, Morrison GM, Morgan R, Reynolds MA. Factors influencing the outcome of regenerative therapy in mandibular Class II furcations: Part I. J Periodontol. 2003 Sep;74(9):1255-68. doi: 10.1902/jop.2003.74.9.1255. PMID 14584858
- [Background] Eickholz P, Horr T, Klein F, Hassfeld S, Kim TS. Radiographic parameters for prognosis of periodontal healing of infrabony defects: two different definitions of defect depth. J Periodontol. 2004 Mar;75(3):399-407. doi: 10.1902/jop.2004.75.3.399. PMID 15088878
- [Background] Crea A, Deli G, Littarru C, Lajolo C, Orgeas GV, Tatakis DN. Intrabony defects, open-flap debridement, and decortication: a randomized clinical trial. J Periodontol. 2014 Jan;85(1):34-42. doi: 10.1902/jop.2013.120753. Epub 2013 Mar 28. PMID 23537123
- [Background] Kiany F, Moloudi F. Amnion membrane as a novel barrier in the treatment of intrabony defects: a controlled clinical trial. Int J Oral Maxillofac Implants. 2015 May-Jun;30(3):639-47. doi: 10.11607/jomi.3590. PMID 26009915
- [Background] Koob TJ, Rennert R, Zabek N, Massee M, Lim JJ, Temenoff JS, Li WW, Gurtner G. Biological properties of dehydrated human amnion/chorion composite graft: implications for chronic wound healing. Int Wound J. 2013 Oct;10(5):493-500. doi: 10.1111/iwj.12140. Epub 2013 Aug 1. PMID 23902526
- [Background] Koob TJ, Lim JJ, Massee M, Zabek N, Rennert R, Gurtner G, Li WW. Angiogenic properties of dehydrated human amnion/chorion allografts: therapeutic potential for soft tissue repair and regeneration. Vasc Cell. 2014 May 1;6:10. doi: 10.1186/2045-824X-6-10. eCollection 2014. PMID 24817999
- [Background] Chakraborthy S, Sambashivaiah S, Kulal R, Bilchodmath S. Amnion and Chorion Allografts in Combination with Coronally Advanced Flap in the Treatment of Gingival Recession: A Clinical Study. J Clin Diagn Res. 2015 Sep;9(9):ZC98-ZC101. doi: 10.7860/JCDR/2015/12971.6572. Epub 2015 Sep 1. PMID 26501023
- [Background] Avila-Ortiz G, De Buitrago JG, Reddy MS. Periodontal regeneration - furcation defects: a systematic review from the AAP Regeneration Workshop. J Periodontol. 2015 Feb;86(2 Suppl):S108-30. doi: 10.1902/jop.2015.130677. PMID 25644295
- [Background] Albandar JM, Brown LJ, Loe H. Clinical features of early-onset periodontitis. J Am Dent Assoc. 1997 Oct;128(10):1393-9. doi: 10.14219/jada.archive.1997.0058. PMID 9332140
- [Background] Genco RJ, Borgnakke WS. Risk factors for periodontal disease. Periodontol 2000. 2013 Jun;62(1):59-94. doi: 10.1111/j.1600-0757.2012.00457.x. PMID 23574464
- [Background] Preshaw PM. Host response modulation in periodontics. Periodontol 2000. 2008;48:92-110. doi: 10.1111/j.1600-0757.2008.00252.x. No abstract available. PMID 18715360
- [Background] Waerhaug J. The infrabony pocket and its relationship to trauma from occlusion and subgingival plaque. J Periodontol. 1979 Jul;50(7):355-65. doi: 10.1902/jop.1979.50.7.355. PMID 381633
- [Background] Laurell L, Gottlow J, Zybutz M, Persson R. Treatment of intrabony defects by different surgical procedures. A literature review. J Periodontol. 1998 Mar;69(3):303-13. doi: 10.1902/jop.1998.69.3.303. PMID 9579616
- [Background] Ivanovic A, Nikou G, Miron RJ, Nikolidakis D, Sculean A. Which biomaterials may promote periodontal regeneration in intrabony periodontal defects? A systematic review of preclinical studies. Quintessence Int. 2014 May;45(5):385-95. doi: 10.3290/j.qi.a31538. PMID 24634903
- [Background] Claffey N, Egelberg J. Clinical characteristics of periodontal sites with probing attachment loss following initial periodontal treatment. J Clin Periodontol. 1994 Nov;21(10):670-9. doi: 10.1111/j.1600-051x.1994.tb00785.x. PMID 7852611

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Test Group
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Test Group
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.53 (15.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 4
Iniital Probing Depth [Mean (Standard Deviation); unit: millimeter] | 7.67 (1.12)
Gingival Recession [Mean (Standard Deviation); unit: millimeter] | 0.44 (1.01)
Clinical Attachement Level [Mean (Standard Deviation); unit: millimeter] | 8.11 (1.62)

OUTCOME MEASURES:

1. Primary Outcome: Probing Depth Change
Description: Probing depth was measured at intrabony defect following surgical procedure.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: millimeter
Arm/Group | Test Group
Number analyzed (Participants) | 4
millimeter | 4.22 (0.73)

2. Primary Outcome: Clinical Attachment Change
Description: Clinical Attachment is defined as the sum of probing depth and gingival recession. The amount of gain of attachment level will be measured.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Test Group
Number analyzed (Participants) | 4
mm | 2.44 (2.24)

ADVERSE EVENTS:
Time Frame: up to 6 months
Arm/Group | Test Group
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-09-10): https://cdn.clinicaltrials.gov/large-docs/76/NCT03095976/Prot_SAP_ICF_000.pdf